CLINICAL TRIAL: NCT00735397
Title: An Open-Label Extension Phase of the Double-Blind, Placebo-Controlled, Dose-Escalation, Parallel-Group Studies to Evaluate the Efficacy and Safety of E2007 (Perampanel) Given as Adjunctive Therapy in Subjects With Refractory Partial Seizures
Brief Title: Evaluation of the Efficacy and Safety of E2007 (Perampanel) Given as Adjunctive Therapy in Subjects With Refractory Partial Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2007-G000-307
Record Dates: First submitted 2008-08-13; First posted 2008-08-14 (Estimated); Results first posted 2016-01-26 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-02

CONDITIONS: Epilepsy
Keywords: Partial onset seizures
MeSH Terms: conditions — Epilepsy | interventions — perampanel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Perampanel (Experimental): Participants previously receiving perampanel/placebo in the double blind-study, were titrated to receive perampanel 2 mg to 12 mg, once daily in the Open-Label Extension (OLE) study up to approximately 5 years.
  Interventions: Drug: perampanel

INTERVENTIONS:
Drug: perampanel — Perampanel 2 mg to 12 mg, once daily in the Open-Label Extension (OLE) study up to approximately 5 years

SUMMARY:
The purpose of this study was to evaluate the safety and tolerability of perampanel (up to 12 mg/day) given as adjunctive treatment in subjects with refractory partial seizures and to evaluate the maintenance of effect of perampanel for the control of refractory partial seizures.

DETAILED DESCRIPTION:
This was an open-label extension (OLE) study for subjects who completed one of the following double-blind, placebo-controlled, Phase 3 studies: E2007-G000-304 (NCT00699972), E2007-G000-305 (NCT00699582), and E2007-G000-306 (NCT00700310). This OLE study consisted of 2 phases: an Open-label Treatment Phase (comprised of a 16-week blinded Conversion Period and a 256-week Maintenance Period) and a Follow-up Phase (4 weeks). During the Conversion Period, subjects and investigators remained blinded to the treatment received in the previous DB study. To achieve this, all subjects continued to take 6 tablets of study medication (2 mg perampanel or matching placebo) or fewer as they were instructed during the core Double-Blind (DB) study. During the open-label Maintenance Period, subjects were treated with the perampanel dose that provided the best combination of individual efficacy and tolerability.

ELIGIBILITY:
Inclusion Criteria:

Each participant who met the following criteria were enrolled in this study:

1. Who completed Visit 8 of study E2007-G000-304, E2007-G000-305, or E2007-G000-306 and complied with the inclusion and exclusion criteria for that study (excluding criteria that are related to seizure occurrences).
2. Provided written informed consent signed by participant or legal guardian prior to entering the study or undergoing any study procedures (If the written informed consent was provided by the legal guardian because the participant was unable to do so, a written or verbal assent from the participant was obtained).
3. Who was considered reliable and willing to be available for the study period and record seizures and report adverse events them self or have a caregiver who can record and report the events for them.
4. Females who were either of non-childbearing potential (defined as having undergone surgical sterilization, or postmenopausal [>age 50 and amenorrheic for 12 months]) or of childbearing potential. Females of childbearing potential were enrolled only if they agreed to be abstinent or continue using at least 1 medically acceptable method of contraception (eg, a double-barrier method [eg, condom + spermicide, condom + diaphragm with spermicide], IUD, or have a vasectomised partner) throughout the study period and for 2 months after the last dose of study drug. Women using hormonal contraceptives were required to use an additional approved method of contraception (as described previously) continuously throughout the entire study period and for 2 months after the last dose of study drug. (It was not required for male subjects to use contraceptive measures based on preclinical toxicology data).
5. Continued to be treated with a stable dose of 1 or a maximum of 3 approved anti-epileptic drugs.

Exclusion Criteria:

Participants who met the following criteria were excluded from the study:

1. Those who, for any reason, discontinued early from the preceding double-blind study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1218 (Actual)
Dates: Start 2008-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Gee, PhD., Study Director — Eisai Limited
Locations (202):
- United States (52):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Fresno, California
  - San Francisco, California
  - Ventura, California
  - Denver, Colorado
  - Fort Collins, Colorado
  - Washington D.C., District of Columbia
  - Gulf Breeze, Florida
  - Jacksonville, Florida
  - Orlando, Florida
  - Tallahassee, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Suwanee, Georgia
  - Boise, Idaho
  - Indianapolis, Indiana
  - Ames, Iowa
  - Lexington, Kentucky
  - Houma, Louisiana
  - Baltimore, Maryland
  - Bethesda, Maryland
  - Hattiesburg, Mississippi
  - Chesterfield, Missouri
  - Kansas City, Missouri
  - St Louis, Missouri
  - Albany, New York
  - Buffalo, New York
  - Great Neck, New York
  - Lawrence, New York
  - New York, New York
  - Rochester, New York
  - Syracuse, New York
  - Asheville, North Carolina
  - Akron, Ohio
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Toledo, Ohio
  - Tulsa, Oklahoma
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Memphis, Tennessee
  - Dallas, Texas
  - El Paso, Texas
  - Houston, Texas
  - Salt Lake City, Utah
  - Richmond, Virginia
  - Seattle, Washington
  - Madison, Wisconsin
- Argentina (9):
  - Buenos Aires
  - Capital Federal
  - Córdoba
  - La Plata, Buenos Aires
  - Lanus Oeste, Buenos Aires
  - Rosario
  - Salta
  - San Miguel de Tucumán
  - Villa Nueva
- Australia (4):
  - Woodville, South Australia
  - Fitzroy, Victoria
  - Heidelberg, Victoria
  - Parkville, Victoria
- Austria (3):
  - Graz
  - Innsbruck
  - Linz
- Belgium (3):
  - Brussels
  - Leuven
  - Ottignies
- Bulgaria (3):
  - Pleven
  - Plovdiv
  - Sofia
- Canada (4):
  - Calgary, Alberta
  - London, Ontario
  - Toronto, Ontario
  - Greenfield Park, Quebec
- Chile (2):
  - Santiago
  - Valdivia
- China (4):
  - Beijing
  - Chengdu
  - Chongqing
  - Shanghai
- Czechia (2):
  - Olomouc
  - Prague
- Estonia (2):
  - Tallinn
  - Tartu
- Finland (2):
  - Kuopio
  - Tampere
- France (5):
  - Béthune
  - Bron
  - Montpellier
  - Rennes
  - Toulouse
- Germany (13):
  - Berlin
  - Bernau
  - Bielefeld
  - Bonn
  - Düsseldorf
  - Erlangen
  - Göttingen
  - Kehl-Kork
  - Mainz
  - Marburg
  - München
  - Ulm
  - Westerstede
- Thessaloniki, Greece
- Hong Kong (4):
  - Hong Kong
  - Kowloon
  - Pokfulam
  - Shatin
- Hungary (2):
  - Budapest
  - Kecskemét
- India (9):
  - Hyderabad
  - Jaipur
  - Mangalore
  - Mumbai
  - Nagpur
  - Nashik
  - New Delhi
  - Pune
  - Visakhapatnam
- Israel (6):
  - Ashkelon
  - Haifa
  - Holon
  - Kfar Saba
  - Petah Tikva
  - Ramat Gan
- Italy (4):
  - Florence
  - Genova
  - Milan
  - Napoli
- Latvia (2):
  - Riga
  - Valmiera
- Lithuania (3):
  - Kaunas
  - Klaipėda
  - Vilnius
- Malaysia (2):
  - Kuala Lumpur
  - Kuala Terengganu
- Mexico (4):
  - Aguascalientes
  - Mexico City, Distrito Federal
  - Monterrey, Nuevo Leon
  - San Luis Potosí City
- Netherlands (2):
  - Heeze
  - Zwolle
- Philippines (2):
  - Ermita
  - Makati City
- Poland (5):
  - Bialystok
  - Gdansk
  - Katowice
  - Lublin
  - Warsaw
- Portugal (3):
  - Coimbra
  - Lisbon
  - Porto
- Bucharest, Romania
- Russia (9):
  - Kazan'
  - Moscow
  - Nizhny Novgorod
  - Omsk
  - Samara
  - Smolensk
  - Tyumen
  - Yaroslavl
  - Yekaterinburg
- Serbia (3):
  - Belgrade
  - Niš
  - Novi Sad
- South Africa (3):
  - Johannesburg, Gauteng
  - Cape Town, Western Cape
  - Cape Town
- South Korea (4):
  - Busan
  - Daegu
  - Pusan
  - Seoul
- Spain (7):
  - Granada, Andalusia
  - Barakaldo, Basque Country
  - Badalona, Catalonia
  - Barcelona, Catalonia
  - Alcorcón, Madrid, Communidad de
  - Madrid, Madrid, Communidad de
  - Valencia, Valencia
- Sweden (2):
  - Gothenburg
  - Linköping
- Taiwan (4):
  - Kaohsiung City
  - Taichung
  - Tainan
  - Taoyuan District
- Thailand (3):
  - Bangkok
  - Chiang Mai
  - Muang
- Ukraine (5):
  - Donetsk
  - Kharkiv
  - Kyiv
  - Lviv
  - Uzhhorod
- United Kingdom (4):
  - Liverpool
  - London
  - Middlesbrough
  - Stoke-on-Trent

REFERENCES:
- [Derived] Maguire M. Response to "Perampanel and pregnancy: Could experience be a gloomy lantern that does not even illuminate its bearer?". Epilepsy Behav. 2022 Apr;129:108654. doi: 10.1016/j.yebeh.2022.108654. Epub 2022 Mar 16. No abstract available. PMID 35305920
- [Derived] Krauss GL, Perucca E, Kwan P, Ben-Menachem E, Wang XF, Shih JJ, Patten A, Yang H, Williams B, Laurenza A. Final safety, tolerability, and seizure outcomes in patients with focal epilepsy treated with adjunctive perampanel for up to 4 years in an open-label extension of phase III randomized trials: Study 307. Epilepsia. 2018 Apr;59(4):866-876. doi: 10.1111/epi.14044. Epub 2018 Mar 25. PMID 29574701
- [Derived] Rosenfeld W, Conry J, Lagae L, Rozentals G, Yang H, Fain R, Williams B, Kumar D, Zhu J, Laurenza A. Efficacy and safety of perampanel in adolescent patients with drug-resistant partial seizures in three double-blind, placebo-controlled, phase III randomized clinical studies and a combined extension study. Eur J Paediatr Neurol. 2015 Jul;19(4):435-45. doi: 10.1016/j.ejpn.2015.02.008. Epub 2015 Mar 5. PMID 25823975
- [Derived] Krauss GL, Perucca E, Ben-Menachem E, Kwan P, Shih JJ, Clement JF, Wang X, Bagul M, Gee M, Zhu J, Squillacote D. Long-term safety of perampanel and seizure outcomes in refractory partial-onset seizures and secondarily generalized seizures: results from phase III extension study 307. Epilepsia. 2014 Jul;55(7):1058-68. doi: 10.1111/epi.12643. Epub 2014 May 27. PMID 24867391

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label Extension (OLE) study for participants who completed one of the following double-blind (DB), placebo-controlled, Phase 3 studies: E2007-G000-304 (NCT00699972), E2007-G000-305(NCT00699582), and E2007-G000-306 (NCT00700310).
Pre-assignment Details: From a total of 1218 participants who provided informed consent, 2 participants were lost to follow-up and did not have any postbaseline safety data after the first OLE dose.
Groups:
- Perampanel: Participants previously receiving perampanel/placebo in the DB study, were titrated to receive perampanel 2 mg to 12 mg, once daily in the OLE study up to approximately 5 years.
Period: Overall Study
Arm/Group | Perampanel
Started | 1218
Completed | 35
Not Completed | 1183
Not completed — Adverse Event | 194
Not completed — Lost to Follow-up | 33
Not completed — Participant choice | 252
Not completed — Inadequate therapeutic effect | 202
Not completed — Administrative/Other | 502

BASELINE CHARACTERISTICS:
Arm/Group | Perampanel
Number analyzed (Participants) | 1218
Age, Continuous [Median (Full Range); unit: years] | 33 [12 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 607
  Male | 611

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Non-Serious Adverse Events (AEs) and Treatment-emergent Serious Adverse Events (SAEs)
Description: An AE was defined as any untoward medical occurrence in a clinical investigation participant administered with an investigational product. A SAE was defined as any untoward medical occurrence that at any dose; resulted in death, was life-threatening (ie, the participant was at immediate risk of death from the AE as it occurred; this did not include an event that, had it occurred in a more severe form or was allowed to continue, might have caused death), required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, or was as a congenital anomaly/birth defect (in the child of a participant who was exposed to the study drug). In this study, treatment emergent AEs (defined as an AE (serious or non-serious) that started/increased in severity on/after the first dose of study medication up to 30 days after the final dose of study medication) were assessed.
Time Frame: From date of first dose of perampanel up to 30 days after the last dose of perampanel or up to approximately 5 years.
Population: The safety analysis set (SAS) was defined as participants who provided informed consent for the OLE study, received at least 1 dose of perampanel in the OLE study, and had at least 1 postdose safety assessment in the OLE study.
Measure: Number; unit: participants
Arm/Group | Perampanel
Number analyzed (Participants) | 1216
participants
  Treatment-emergent non serious AEs | 1018
  Treatment-emergent SAEs | 288

2. Secondary Outcome: Median Percent Change in Seizure Frequency Per 28 Days Relative to Pre-Perampanel Baseline.
Description: Seizure frequency was derived from information (seizure count and type) recorded in participant diary. The seizure frequency per 28 days was calculated as the number of seizures divided by the number of days in the interval and multiplied by 28. The percent change in 28-day seizure frequency from pre-perampanel baseline was assessed for all partial-onset seizure types. The pre-perampanel baseline was defined as: (1) for participants who had been assigned to placebo treatment in the core DB study, the pre-perampanel baseline was computed from all data during the core DB study, and (2) for participants who had been assigned to perampanel in the core DB study, the pre-perampanel baseline was computed from the pre-randomization phase of the core DB study.
Time Frame: Pre-perampanel Baseline and Weeks (1-13, 14-26, 27-39, 40-52, 53-65, 66-78, 79-91, 92-104, 105-117, 118-130, 131-143, 144-156, 157-169, 170-182, 183-195, 196-208, 209-221, 222-234, 235-247, and 248-260)
Population: Full Intent-to-treat population (ITT), defined as participants who provided informed consent for the OLE, received at least 1 dose of perampanel in the OLE, and had valid seizure data for overall, Complex Partial Plus Secondarily Generalized Seizures and Secondarily Generalized Seizures arm, respectively during the perampanel treatment duration.
Measure: Median (Full Range); unit: Percent change
Groups:
- Overall; Complex Partial Plus Secondarily Generalized Seizures; Secondarily Generalized Seizures: Participants previously receiving perampanel/placebo in the DB study, were titrated to receive perampanel 2 mg to 12 mg, once daily in the OLE study up to approximately 5 years.
Arm/Group | Overall | Complex Partial Plus Secondarily Generalized Seizures | Secondarily Generalized Seizures
Number analyzed (Participants) | 1217 | 1126 | 510
Percent change
  Weeks 1-13 | -29.14 [-100.0 to 737.1] | -32.42 [-100.0 to 14858.2] | -54.95 [-100.0 to 530.8]
  Weeks 14-26, n = 1159, 1073, 482 | -38.54 [-100.0 to 866.6] | -43.19 [-100.0 to 12965.9] | -65.69 [-100.0 to 628.6]
  Wekks 27-39, n = 1088, 1011, 458 | -42.81 [-100.0 to 780.6] | -46.22 [-100.0 to 14092.3] | -77.47 [-100.0 to 756.0]
  Weeks 40-52, n = 969, 903, 416 | -46.22 [-100.0 to 685.7] | -49.39 [-100.0 to 898.1] | -81.15 [-100.0 to 898.1]
  Weeks 53-65, n = 882, 819, 381 | -49.34 [-100.0 to 526.4] | -54.95 [-100.0 to 1071.4] | -80.69 [-100.0 to 891.2]
  Weeks 66-78, n = 822, 762, 357 | -51.65 [-100.0 to 861.5] | -56.25 [-100.0 to 620.9] | -79.98 [-100.0 to 891.2]
  Weeks 79-91, n = 762, 703, 329 | -53.06 [-100.0 to 697.5] | -55.38 [-100.0 to 1000.6] | -90.68 [-100.0 to 1071.4]
  Weeks 92-104, n = 720, 664, 313 | -56.59 [-100.0 to 660.9] | -62.11 [-100.0 to 717.2] | -90.33 [-100.0 to 891.2]
  Weeks 105-117, n = 676, 624, 295 | -59.07 [-100.0 to 627.9] | -63.62 [-100.0 to 627.9] | -84.98 [-100.0 to 1071.4]
  Weeks 118-130, n = 642, 590, 279 | -60.89 [-100.0 to 540.0] | -66.75 [-100.0 to 821.1] | -100.00 [-100.0 to 1281.0]
  Weeks 131-143, n = 583, 535, 258 | -60.67 [-100.0 to 716.0] | -65.46 [-100.0 to 717.5] | -99.70 [-100.0 to 801.1]
  Weeks 144-156, n = 517, 478, 231 | -61.45 [-100.0 to 570.2] | -67.95 [-100.0 to 562.6] | -100.00 [-100.0 to 936.3]
  Weeks 157-169, n = 429, 396, 187 | -65.46 [-100.0 to 418.3] | -72.21 [-100.0 to 264.4] | -100.00 [-100.0 to 350.0]
  Weeks 170-182, n = 323, 297, 137 | -64.29 [-100.0 to 367.4] | -76.37 [-100.0 to 268.2] | -100.00 [-100.0 to 269.2]
  Weeks 183-195, n = 210, 193, 89 | -66.63 [-100.0 to 698.7] | -74.78 [-100.0 to 867.1] | -100.00 [-100.0 to 320.3]
  Weeks 196-208, n = 119, 111, 47 | -73.30 [-100.0 to 671.8] | -80.77 [-100.0 to 671.8] | -100.00 [-100.0 to 147.3]
  Weeks 209-221, n = 59, 57, 22 | -72.47 [-100.0 to 226.4] | -80.69 [-100.0 to 211.4] | -100.00 [-100.0 to 55.8]
  Weeks 222-234, n = 37, 36, 11 | -81.36 [-100.0 to 175.3] | -89.02 [-100.0 to 75.3] | -99.11 [-100.0 to 75.3]
  Weeks 235-247, n = 14, 13, 2 | -78.10 [-100.0 to 200.4] | -100.0 [-100.0 to 71.4] | -100.00 [-100.0 to -100.0]
  Weeks 248-260, n = 5, 5, 1 | -97.16 [-100.0 to 250.4] | -98.39 [-100.0 to -90.0] | -98.39 [-98.39 to -98.39]

3. Secondary Outcome: Percentage of Participants Who Experienced a 50% or Greater Reduction in Seizure Frequency Per 28 Days Relative to the Pre-Perampanel Baseline.
Description: Seizure frequency was derived from information (seizure count and type) recorded in participant diary. The percentage of participants who experienced a 50% or greater reduction in seizure frequency per 28 days relative to the pre-perampanel Baseline(responders) was assessed. The pre-perampanel baseline was defined as: (1) for participants who had been assigned to placebo treatment in the core DB study, the Pre-perampanel baseline was computed from all data during the core Double-Blind (DB) study, and (2) for participants who had been assigned to perampanel in the core DB study, the pre-perampanel baseline was computed from the pre-randomization phase of the core DB study. The data is presented as percent responders.
Time Frame: Pre-perampanel Baseline and Weeks (1-13, 14-26, 27-39, 40-52, 53-65, 66-78, 79-91, 92-104, 105-117, 118-130, 131-143, 144-156, 157-169, 170-182, 183-195, 196-208, 209-221, 222-234, 235-247, 248-260)
Population: as for outcome 2
Measure: Number; unit: Percent responders
Arm/Group | Overall | Complex Partial Plus Secondarily Generalized Seizures | Secondarily Generalized Seizures
Number analyzed (Participants) | 1217 | 1126 | 510
Percent responders
  Weeks 1-13 | 30.8 | 34.8 | 54.5
  Weeks 14-26, n = 1159, 1073, 482 | 40.9 | 43.4 | 58.7
  Weeks 27-39, n = 1088, 1011, 458 | 44.2 | 47.3 | 63.3
  Weeks 40-52, n = 969, 903, 416 | 45.6 | 49.4 | 67.8
  Weeks 53-65, n = 882, 819, 381 | 49.5 | 53.2 | 65.6
  Weeks 66-78, n = 822, 762, 357 | 51.5 | 54.9 | 66.1
  Weeks 79-91, n = 762, 703, 329 | 52.9 | 55.6 | 66.0
  Weeks 92-104, n = 720, 664, 313 | 57.2 | 58.6 | 69.3
  Weeks 105-117, n = 676, 624, 295 | 57.1 | 59.5 | 68.1
  Weeks 118-130, n = 642, 590, 279 | 58.9 | 61.9 | 71.3
  Weeks 131-143, n = 583, 535, 258 | 59.3 | 61.5 | 71.3
  Weeks 144-156, n = 517, 478, 231 | 60.9 | 62.6 | 74.0
  Weeks 157-169, n = 429, 396, 187 | 63.2 | 65.7 | 76.5
  Weeks 170-182, n = 323, 297, 137 | 60.1 | 64.3 | 78.8
  Weeks 183-195, n = 210, 193, 89 | 62.9 | 68.4 | 80.9
  Weeks 196-208, n = 119, 111, 47 | 64.7 | 71.2 | 85.1
  Weeks 209-221, n = 59, 57, 22 | 67.8 | 73.7 | 77.3
  Weeks 222-234, n = 37, 36, 11 | 73.0 | 75.0 | 72.7
  Weeks 235-247, n = 14, 13, 2 | 64.3 | 69.2 | 100.0
  Weeks 248-260, n = 5, 5, 1 | 80.0 | 100.0 | 100.0

ADVERSE EVENTS:
Time Frame: From date of first dose of perampanel up to 30 days after the last dose of perampanel or up to approximately 5 years
Description: In this study, treatment emergent AE (defined as an AE/SAE that started/increased in severity on/after the first dose of study medication up to 30 days after the final dose of study medication) were assessed.
Arm/Group | Perampanel
Serious Adverse Events (participants affected / at risk) | 288/1216
Other Adverse Events (participants affected / at risk) | 1018/1216
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Perampanel (N=1216)
Hypertension (Vascular disorders) | 2
Aortic aneurysm (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Abortion induced (Surgical and medical procedures) | 6
Medical device removal (Surgical and medical procedures) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2
Abortion spontaneous incomplete (Pregnancy, puerperium and perinatal conditions) | 1
Gait disturbance (General disorders) | 2
Pain (General disorders) | 2
Cyst (General disorders) | 1
Death (General disorders) | 1
Drug ineffective (General disorders) | 1
Fatigue (General disorders) | 1
General physical health deterioration (General disorders) | 1
Hyperthermia (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pyrexia (General disorders) | 1
Sudden death (General disorders) | 1
Aggression (Psychiatric disorders) | 14
Psychotic disorder (Psychiatric disorders) | 8
Suicidal ideation (Psychiatric disorders) | 6
Affective disorder (Psychiatric disorders) | 5
Depression (Psychiatric disorders) | 5
Acute psychosis (Psychiatric disorders) | 4
Suicide attempt (Psychiatric disorders) | 4
Disorientation (Psychiatric disorders) | 3
Paranoia (Psychiatric disorders) | 3
Abnormal behaviour (Psychiatric disorders) | 2
Agitation (Psychiatric disorders) | 2
Adjustment disorder (Psychiatric disorders) | 1
Anger (Psychiatric disorders) | 1
Catanoia (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Delusion (Psychiatric disorders) | 1
Delusion of grandeur (Psychiatric disorders) | 1
Epileptic psychosis (Psychiatric disorders) | 1
Hallucination,auditory (Psychiatric disorders) | 1
Homicidal ideation (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Irritability (Psychiatric disorders) | 1
Major depression (Psychiatric disorders) | 1
Mental disorder due to a general medical condition (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Mood altered (Psychiatric disorders) | 1
Negativism (Psychiatric disorders) | 1
Obsessive thoughts (Psychiatric disorders) | 1
Personlaity change due to a general medical condition (Psychiatric disorders) | 1
Postictal psychosis (Psychiatric disorders) | 1
Dysfuntional uterine bleeding (Reproductive system and breast disorders) | 2
Bartholinitis (Reproductive system and breast disorders) | 1
Breast enlargement (Reproductive system and breast disorders) | 1
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1
Menstrual disorder (Reproductive system and breast disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
Ovarian mass (Reproductive system and breast disorders) | 1
Ovarian rupture (Reproductive system and breast disorders) | 1
Polycystic ovaries (Reproductive system and breast disorders) | 1
Uterine cyst (Reproductive system and breast disorders) | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 1
Uterine polyp (Reproductive system and breast disorders) | 1
Head injury (Injury, poisoning and procedural complications) | 12
Ankle fracture (Injury, poisoning and procedural complications) | 7
Fall (Injury, poisoning and procedural complications) | 5
Road traffic accident (Injury, poisoning and procedural complications) | 5
Toxicity to various agents (Injury, poisoning and procedural complications) | 5
Contusion (Injury, poisoning and procedural complications) | 4
Facial bones fracture (Injury, poisoning and procedural complications) | 4
Craniocerebral injury (Injury, poisoning and procedural complications) | 3
Foot fracture (Injury, poisoning and procedural complications) | 3
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 3
Accidental overdose (Injury, poisoning and procedural complications) | 2
Brain contusion (Injury, poisoning and procedural complications) | 2
Clavicle fracture (Injury, poisoning and procedural complications) | 2
Extradural haematoma (Injury, poisoning and procedural complications) | 2
Fibula fracture (Injury, poisoning and procedural complications) | 2
Hand fracture (Injury, poisoning and procedural complications) | 2
Humerus fracture (Injury, poisoning and procedural complications) | 2
Jaw fracture (Injury, poisoning and procedural complications) | 2
Laceration (Injury, poisoning and procedural complications) | 2
Lower limb fracture (Injury, poisoning and procedural complications) | 2
Rib fracture (Injury, poisoning and procedural complications) | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 2
Tibia fracture (Injury, poisoning and procedural complications) | 2
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 2
Abdominal injury (Injury, poisoning and procedural complications) | 1
Animal bite (Injury, poisoning and procedural complications) | 1
Burns second degree (Injury, poisoning and procedural complications) | 1
Burns third degree (Injury, poisoning and procedural complications) | 1
Cartilage injury (Injury, poisoning and procedural complications) | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1
Concussion (Injury, poisoning and procedural complications) | 1
Epidural haemorrhage (Injury, poisoning and procedural complications) | 1
Excoriation (Injury, poisoning and procedural complications) | 1
Forearm fracture (Injury, poisoning and procedural complications) | 1
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Intentional overdose (Injury, poisoning and procedural complications) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1
Muscle strain (Injury, poisoning and procedural complications) | 1
Neck injury (Injury, poisoning and procedural complications) | 1
Post concussion syndrome (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Skin laceration (Injury, poisoning and procedural complications) | 1
Skull fracture (Injury, poisoning and procedural complications) | 1
Skull fractured base (Injury, poisoning and procedural complications) | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1
Traumatic iritis (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Clostridium test positive (Investigations) | 1
Heart rate irregular (Investigations) | 1
Weight decreased (Investigations) | 1
Angina pectoris (Cardiac disorders) | 3
Atrial fibrillation (Cardiac disorders) | 3
Bradycardia (Cardiac disorders) | 2
Acute coronary syndrome (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Atrioventricular dissociation (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardiovascular insufficiency (Cardiac disorders) | 1
Coronary artery stenosis (Cardiac disorders) | 1
Mitral valve incompetence (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Sick sinas syndrome (Cardiac disorders) | 1
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 1
Skull malformation (Congenital, familial and genetic disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Convulsion (Nervous system disorders) | 43
Status epilepticus (Nervous system disorders) | 16
Epilepsy (Nervous system disorders) | 15
Dizziness (Nervous system disorders) | 6
Grand mal convulsion (Nervous system disorders) | 6
Seizure cluster (Nervous system disorders) | 6
Ataxia (Nervous system disorders) | 3
Partial seizures (Nervous system disorders) | 3
Partial seizures with secondary generalisation (Nervous system disorders) | 3
Cerebral haemorrhage (Nervous system disorders) | 2
Cerebrovascular accident (Nervous system disorders) | 2
Drug withdrawal convulsions (Nervous system disorders) | 2
Dysarthria (Nervous system disorders) | 2
Hemiparesis (Nervous system disorders) | 2
Hypoasthesia (Nervous system disorders) | 2
Somnolence (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 2
Carotid artery dissection (Nervous system disorders) | 1
Carpal tunnel syndrome (Nervous system disorders) | 1
Central nervous system lesion (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Cognitive disorder (Nervous system disorders) | 1
Coma (Nervous system disorders) | 1
Complex partial seizures (Nervous system disorders) | 1
Dementia Alzheimer's type (Nervous system disorders) | 1
Haemorrhage intracranial (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Incoherent (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Multifocal motor nueropathy (Nervous system disorders) | 1
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1
Postictal paralysis (Nervous system disorders) | 1
Psychomotor hyperactivity (Nervous system disorders) | 1
Simple partial seizures (Nervous system disorders) | 1
Speech disorder (Nervous system disorders) | 1
Spinal cord compression (Nervous system disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1
Temporal lobe epilepsy (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Vertebral artery dissection (Nervous system disorders) | 1
Stupor (Nervous system disorders) | 1
Conjunctivitis allergic (Eye disorders) | 1
Iritis (Eye disorders) | 1
Visual impairment (Eye disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Conductive deafness (Ear and labyrinth disorders) | 1
Gastritis (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 3
Colitis (Gastrointestinal disorders) | 1
Colitis ischaemic (Gastrointestinal disorders) | 1
Colitis microscopic (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Duodenitis (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Small intestine obstruction (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 2
Urinary retention (Renal and urinary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 4
Cholecystitis (Hepatobiliary disorders) | 2
osteoarthritis (Musculoskeletal and connective tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 1
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1
Goitre (Endocrine disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1
Hypochloraemia (Metabolism and nutrition disorders) | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1
Pneumonia (Infections and infestations) | 13
Urinary tract infection (Infections and infestations) | 6
Appendicitis (Infections and infestations) | 5
Device related infection (Infections and infestations) | 2
Postoperative wound infection (Infections and infestations) | 2
Tooth abscess (Infections and infestations) | 2
Wound infection staphylococcal (Infections and infestations) | 2
Abscess limb (Infections and infestations) | 1
Appendicitis perforated (Infections and infestations) | 1
Bacterial disease carrier (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Klebsiella infection (Infections and infestations) | 1
Meningitis (Infections and infestations) | 1
Oral infection (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Post procedural pneumonia (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Renal cyst infection (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Tuberculosis (Infections and infestations) | 1
Typhoid fever (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Perampanel (N=1216)
Fall (Injury, poisoning and procedural complications) | 116
Laceration (Injury, poisoning and procedural complications) | 67
Weight increased (Investigations) | 161
Ataxia (Nervous system disorders) | 84
Balance disorder (Nervous system disorders) | 74
Convulsion (Nervous system disorders) | 78
Dizziness (Nervous system disorders) | 591
Dysarthria (Nervous system disorders) | 61
Headache (Nervous system disorders) | 246
Somnolence (Nervous system disorders) | 266
Diplopia (Eye disorders) | 64
Fatigue (General disorders) | 182
Irritability (General disorders) | 69
Gait disturbacne (General disorders) | 80
Pyrexia (General disorders) | 79
Vertigo (Ear and labyrinth disorders) | 78
Anxiety (Psychiatric disorders) | 79
Depression (Psychiatric disorders) | 82
Insomnia (Psychiatric disorders) | 86
Irritability (Psychiatric disorders) | 125
Diarrhoea (Gastrointestinal disorders) | 84
Nausea (Gastrointestinal disorders) | 115
Vomiting (Gastrointestinal disorders) | 95
Influenza (Infections and infestations) | 70
Nasopharyngitis (Infections and infestations) | 142
Upper respiratory tract infection (Infections and infestations) | 107
Back pain (Musculoskeletal and connective tissue disorders) | 86

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other